CLINICAL TRIAL: NCT02782416
Title: A Randomized Study for Screening Latent Tuberculosis Infection and Observing Preventive Therapy in Patients Preparing for Kidney Transplantation
Brief Title: Screening Latent Tuberculosis Infection and Observing Preventive Therapy in Kidney Transplantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 201309056RINC
Record Dates: First submitted 2016-05-11; First posted 2016-05-25 (Estimated); Last update posted 2016-12-15 (Estimated); Status verified 2016-12

CONDITIONS: Kidney Transplantation
Keywords: Renal; Latent; Tuberculosis
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Waiting for renal transplant_no screening of LTBI (No Intervention): patients with renal failure and are waiting for renal transplant We do routine examination but no LTBI check
- Not waiting for renal transplant (Placebo Comparator): Dialysis patients who are not waiting for renal transplant
  Interventions: Other: Examination of latent tuberculosis
- Status post renal transplant (Other): patients who have received renal transplant
  Interventions: Other: Examination of latent tuberculosis
- Waiting for renal transplant_ screening of LTBI (Experimental): patients with renal failure and are waiting for renal transplant We do routine examination in addition to LTBI check
  Interventions: Other: Examination of latent tuberculosis

INTERVENTIONS:
Other: Examination of latent tuberculosis
  Arms: Not waiting for renal transplant; Status post renal transplant; Waiting for renal transplant_ screening of LTBI

SUMMARY:
Study the prevalence of LTBI in patients who are waiting renal transplant and monitor the incidence of active TB

DETAILED DESCRIPTION:
Study the prevalence of LTBI in patients who are waiting renal transplant and monitor the incidence of active TB

ELIGIBILITY:
Inclusion Criteria:

1. Age between 20-65 and match one of below
2. Waiting renal transplant or status post renal transplant
3. Receiving long term dialysis

Exclusion Criteria:

1. Not agree to be enrolled
2. Suspected active TB
3. HIV patients
4. Viral hepatitis
5. Using immunosuppressants within 3 months before enrollment
6. Receiving lymphokine therapy
7. Hemoglobin < 8 g/dL
8. Serum bilirubin > 2.5 mg/dL
9. AST or ALT > 2 times of upper normal limit
10. Lactation or pregnancy

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2014-01; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
percentage of active TB | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Chin-Chung Shu, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No